CLINICAL TRIAL: NCT01583452
Title: Use of Chewing Gum to Reduce Postoperative Ileus in Pediatric Patients After Gastrointestinal Surgery
Brief Title: Chewing Gum Use to Reduce Post-operative Ileus in Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Gabriela López Jaimez, Pediatrics Resident, Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UGoMaRIPO
Record Dates: First submitted 2012-04-03; First posted 2012-04-24 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Post Operative Ileus
Keywords: Post operative ileus; Gastrointestinal surgery; Chewing gum
MeSH Terms: interventions — Chewing Gum; Forkhead Box Protein M1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chewing Gum Group (Experimental): Group of patients given chewing gum as part of the treatment for prevention of post-operative ileus right after surgery, besides the standard pharmacologic treatment and post-operative care.
  Interventions: Other: Chewing Gum
- No intervention (No Intervention): By observing the clinical evolution of the participants not given chewing gum as a prevention for post-operative ileus, and just given the standard pharmacologic treatment and post-operative care.

INTERVENTIONS:
Other: Chewing Gum — The use of chewing gum as a preventive measure for post-operative ileus
  Other Names: Sugarless chewing gum; Trident; Orbit; Ice Breakers; Smint
  Arms: Chewing Gum Group

SUMMARY:
Post- operative ileus refers to the time after surgery before coordinated electromotor bowel function resumes. It's treatment and prevention may signify an elevated hospitalization cost and the exposure to the patient to adverse effects of drugs.

The current clinical trial has as primary objective to prove the efficacy of chewing gum as a preventive measure of post-operative ileus in pediatric patients after gastrointestinal surgery through the determination of the time the patient takes to tolerate oral intake, pass flatus, present bowel movements and the time of hospital stay.

Patients will be assigned either to the case group (chewing gum + standard treatment) or to the control group (standard treatment), in both of them time from the end of surgery to the moment the patient presents first bowel movement, passes flatus, tolerates oral intake (any type of food) and is discharged from hospital; will be measured in hours and then analyzed to determine the validity of these data.

DETAILED DESCRIPTION:
Postoperative ileus is a relatively common condition seen in patients with gastrointestinal diseases requiring surgery. Treatment and prevention of this condition involves the use of several drugs and devices which increase the length of hospital stay, costs of treatment and morbidity.

In the last years there have been several reports about the use of chewing gum as a preventive measure of postoperative ileus with positive results in the adult population. Most of these studies involve patients who underwent colectomy. In the bibliographic review the investigators found just one study developed specifically with pediatric patients. Results are very similar between the studies; time to present first bowel movement, pass flatus and tolerate oral intake is decreased with statistically significant evidence, meanwhile, the length of hospital stay has been proved to be shortened in just a few studies.

The primary objective in the investigators study is to demonstrate chewing gum can be a cheap and easy therapeutic strategy to reduce the length of hospital stay, by diminishing the incidence and time of postoperative ileus (by the determination of the time patients take to tolerate oral intake, pass flatus and present bowel movements).

The investigators study hypothesis is stated as follows: Use of chewing gum in pediatric patients after gastrointestinal surgery reduces the risk of post-operative ileus by decreasing the time the patient takes to tolerate oral intake, pass flatus and present bowel movements.

Study Design

* Randomized Clinical Trial
* Prospective
* Experimental

Patients will be assigned either to the case group (chewing gum + standard treatment) or to the control group (standard treatment), in both of them time from the end of surgery to the moment the patient presents first bowel movement, passes flatus, tolerates oral intake (any type of food) and is discharged from hospital; will be measured in hours and then analyzed to determine the validity of these data.

Investigators will register any adverse effect related with the use of chewing gum such as: abdominal distension, abdominal pain, nausea, vomiting, ingestion of chewing gum, intestinal obstruction, or any other patient's complain while being in hospital. Medications used during treatment will also be reported with every patient included in the protocol.

There will be no intervention of any pharmaceutic industry or support of any chewing gum brand. Costs of the study will be covered by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who underwent any type of gastrointestinal surgery.

Exclusion Criteria:

* Patients unable to chew
* Patients unable to swallow
* Patients whose clinical status is critical
* Patients with gastrointestinal motility disorders not associated with GI surgeries.
* Patients unable to follow directions about the use of chewing gum

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Lopez, MD, Principal Investigator — Instituto Tecnologico y de Estudios Superiores de Monterey
Locations (1):
- Hospital San Jose Tec de Monterrey, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Vasquez W, Hernandez AV, Garcia-Sabrido JL. Is gum chewing useful for ileus after elective colorectal surgery? A systematic review and meta-analysis of randomized clinical trials. J Gastrointest Surg. 2009 Apr;13(4):649-56. doi: 10.1007/s11605-008-0756-8. Epub 2008 Dec 3. PMID 19050983
- [Background] Johnson MD, Walsh RM. Current therapies to shorten postoperative ileus. Cleve Clin J Med. 2009 Nov;76(11):641-8. doi: 10.3949/ccjm.76a.09051. PMID 19884293
- [Background] Purkayastha S, Tilney HS, Darzi AW, Tekkis PP. Meta-analysis of randomized studies evaluating chewing gum to enhance postoperative recovery following colectomy. Arch Surg. 2008 Aug;143(8):788-93. doi: 10.1001/archsurg.143.8.788. PMID 18711040
- [Background] de Castro SM, van den Esschert JW, van Heek NT, Dalhuisen S, Koelemay MJ, Busch OR, Gouma DJ. A systematic review of the efficacy of gum chewing for the amelioration of postoperative ileus. Dig Surg. 2008;25(1):39-45. doi: 10.1159/000117822. Epub 2008 Feb 21. PMID 18292660
- [Background] Noble EJ, Harris R, Hosie KB, Thomas S, Lewis SJ. Gum chewing reduces postoperative ileus? A systematic review and meta-analysis. Int J Surg. 2009 Apr;7(2):100-5. doi: 10.1016/j.ijsu.2009.01.006. Epub 2009 Jan 31. PMID 19261555
- [Background] Fitzgerald JE, Ahmed I. Systematic review and meta-analysis of chewing-gum therapy in the reduction of postoperative paralytic ileus following gastrointestinal surgery. World J Surg. 2009 Dec;33(12):2557-66. doi: 10.1007/s00268-009-0104-5. PMID 19763686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our study included 5-18 years old patients with gastrointestinal surgery from two institutions (Hospital San José Tec de Monterrey and Hospital Regional Materno Infantil); during April to August 2012. However, because the most common diagnosis in this group of age was appendicitis, only patients with this condition were included at the end.
Pre-assignment Details: Initially our study was focused on patients who had gastrointestinal surgery, however, the main diagnosis of our population of interest was appendicitis; and those children with other diagnosis did not meet the criteria for including them in the study. This way, our final population was children who underwent open or laparoscopic appendectomy.
Groups:
- Chewing Gum Group: Group of patients given chewing gum as part of the treatment for prevention of post-operative ileus right after surgery, plus the standard pharmacologic treatment and post-operative care.
  Chewing Gum: The use of chewing gum as a preventive measure for post-operative ileus
Period: Overall Study
Arm/Group | Chewing Gum Group | No Intervention
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Intervention: By observing the clinical evolution of the participants not given chewing gum as prevention for post-operative ileus, and just given the standard pharmacologic treatment and post-operative care.
- Total: Total of all reporting groups
Arm/Group | Chewing Gum Group | No Intervention | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 9.5 [7.5 to 12] | 8.6 [6 to 11.5] | 9.2 [6 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  Mexico | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Hospital Stay
Description: The time between the end of surgery and hospital discharge, measured in hours
Time Frame: End of surgery to hospital discharge (from 4 to 7 days)
Population: Patients who underwent open or laparoscopic appendectomy and received chewing gum plus standard pharmacologic care, or just pharmacologic care (control group), as a measure to prevent post-operative ileus.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Chewing Gum Group: The time between the end of the surgery and the discharge of the patients, measured in hours.
- Control Group: The time between the end of surgery and the discharge of the patient measured in hours.
Arm/Group | Chewing Gum Group | Control Group
Number analyzed (Participants) | 21 | 20
hours | 79.93 (50.76) | 72.94 (28.33)
Statistical Analysis 1: Comparison: Chewing Gum Group vs Control Group; With a confidence interval of 95%, an alpha risk of 5% and a desired power of 80%; expecting a 24hrs difference between the intervention and the control group, we estimated 20 patients for each one of them; Test type: Superiority or Other; p = 0.665, Kaplan-Meier survival analysis

2. Secondary Outcome: Time to First Flatus
Description: The time between the end of surgery and the moment in which the patient passes first flatus
Time Frame: End of surgery to first flatus (from 1 to 3 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Chewing Gum Group | No Intervention
Number analyzed (Participants) | 21 | 20
hours | 17.18 (8.18) | 24.37 (1.53)
Statistical Analysis 1: Comparison: Chewing Gum Group vs No Intervention; Test type: Superiority or Other; p = 0.094, Kaplan-Meier survival analysis

3. Secondary Outcome: Time to First Bowel Movement
Description: The time between the end of surgery and the moment in which the patient presents first bowel movement.
Time Frame: End of surgery to first bowel motion (from 1 to 7 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Chewing Gum Group | No Intervention
Number analyzed (Participants) | 21 | 20
hours | 29.91 (21.27) | 34.5 (22.78)
Statistical Analysis 1: Comparison: Chewing Gum Group vs No Intervention; Test type: Superiority or Other; p = 0.059, Kaplan-Meier survival analysis

4. Secondary Outcome: Time to Tolerate Feedings (Oral Intake)
Description: The time between the end of surgery to the moment in which the patient can tolerate the intake of fluids or any type of food.
Time Frame: End of surgery to oral intake tolerance (from 1 to 3 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Chewing Gum Group | No Intervention
Number analyzed (Participants) | 21 | 20
hours | 31.21 (25.46) | 27.04 (15.51)
Statistical Analysis 1: Comparison: Chewing Gum Group vs No Intervention; Test type: Superiority or Other; p = 0.830, Kaplan-Meier survival analysis

ADVERSE EVENTS:
Time Frame: During the 5 months in which data was collected
Description: One patient accidentally swallowed the gum without any clinical signs or complications, however with risk of intestinal obstruction.
Arm/Group | Chewing Gum Group | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chewing Gum Group (N=21) | No Intervention (N=20)
Swallowing of chewing gum (Gastrointestinal disorders) | 1 (1) | 0 (0) — One of the patients in the intervention group accidentally swallowed the gum without any clinical implications, however with risk of intestinal obstruction

LIMITATIONS AND CAVEATS:
We had a small number of participants because of time limitations. We included only patients with diagnosis of appendicitis and post-op appendectomy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No